CLINICAL TRIAL: NCT00297284
Title: Pilot and Feasibility Study of Modafinil Treatment to Improve Cognitive Efficiency in SLE Patients
Brief Title: Memory and Attention Problems in Lupus: New Treatment Trial With Modafinil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25085
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2006-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; cognitive efficiency; cognitive dysfunction; cognition; memory; attention; modafinil; provigil
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Cognitive Dysfunction | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
This study is being conducted in order to determine if the FDA-approved drug Modafinil can improve cognitive function in patients with lupus. Modafinil is currently being used to treat excessive sleepiness caused by certain sleep disorders. It has also been shown to improve attention and concentration in some people who don't have lupus or sleep disorders. This study hopes to determine if Modafinil can be used safely and effectively in lupus patients, and improve their quality of life. No medications currently exist for the treatment of lupus-associated cognitive dysfunction.

DETAILED DESCRIPTION:
This is a 6-week pilot and feasibility single-arm, open-label trial of modafinil 200mg orally every morning to improve cognitive efficiency in systemic lupus patients with cognitive difficulties in daily life.

Cognitive dysfunction is a well-recognized manifestation of systemic lupus erythematosus (SLE) whose reported prevalence ranges from 12-87%. SLE-associated cognitive dysfunction often occurs in the absence of frank neuropsychiatric disease (e.g., stroke, depression, psychosis, cerebral vasculitis), medications known to have central nervous system effects, or increased disease activity or flare. Studies of SLE antibodies (most notably the antiphospholipid antibodies) have provided conflicting results with respect to their association with SLE-associated cognitive dysfunction. Thus, despite numerous investigations, the etiology of SLE-associated cognitive dysfunction remains unclear. There is no known means for preventing cognitive dysfunction in SLE. Similarly there are no established or proven treatments for cognitive dysfunction in SLE.

Regardless of its cause, course, or long-term consequences, cognitive dysfunction in SLE is a major cause of distress, compromised performance of everyday activities, and decreased quality of life. Thus, treatment of decreased cognitive performance in SLE when it occurs, no matter how mild, and regardless of its potential for permanence or progression, is of paramount importance. It is imperative to provide SLE patients with cognitive performance difficulties with the means to functionally cope with their impairments so that they can maintain, if not regain their independence.

Modafinil is a safe, orally administered wakefulness-promoting agent approved for use in adults suffering from narcolepsy, idiopathic hypersomnia, obstructive sleep apnea, and shift work sleep syndrome. Since its FDA approval, it has been used for many additional varied conditions including depression, fatigue, fibromyalgia, myotonic dystrophy, organic brain syndrome, sleep deprivation, Parkinson's, and drug-induced somnolence. It has also been used in helicopter and airplane pilots to enhance their attentiveness during long flights. Some of our SLE patients have been prescribed modafinil for narcolepsy or associated fatigue.

Modafinil has broad efficacy in health and illness. It enhances cognitive function in normal young adult males, as tested by digit span, visual pattern recognition memory, spatial planning and stop-signal reaction time. While the majority of patients prescribed modafinil received the drug for non-cognitive indications (e.g., fatigue, sleepiness), several have reported improved cognitive function, especially with respect to tasks that require attention and concentration.

We hypothesize that Modafinil, an FDA-approved, non-specific wakefulness-promoting agent with minimal side effects, is safe and effective when used to improve cognitive efficiency in SLE patients who identify cognitive dysfunction in themselves.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill ACR Classification Criteria for SLE
* >18 and < 60 years old
* English-speaking/reading
* Has a treating rheumatologist at the Hospital for Special Surgery
* Estimated premorbid verbal I.Q. >80 measured by the North American Adult Reading Test
* Functional difficulties due to cognitive dysfunction defined as positive endorsement of ≥6 items on the Cognitive Symptoms Inventory (CSI). The CSI is a 21-item, self-report questionnaire designed to assess ability to perform everyday activities in patients with rheumatic disease.47
* No physical or mental disabilities that would preclude or confound the results of the neuropsychological testing, e.g., compromised use of hands, severe visual or hearing impairment
* Able to read normal newsprint and hear a normal speaking voice
* Normotensive at time of enrollment with or without medication
* No arrhythmia or left ventricular hypertrophy on ECG
* Adequate contraception (barrier method)

Exclusion Criteria:

* Global cognitive impairment as measured by a Modified Mini Mental Status<77
* History of arrhythmia; known history of left ventricular hypertrophy, mitral valve prolapse with syndrome, or other significant cardiovascular disease with a reduced ejection fraction
* Renal insufficiency (creatinine clearance < 30 ml/min) including dialysis patients
* Known liver disease (e.g., active hepatitis) or any liver function test >2x upper limit of normal (transaminases or GGTP)
* Significant and serious SLE activity defined as active central nervous system disease, active nephritis, ulcerative skin disease. Other active SLE-associated conditions involving major organ systems may be excluded at the discretion of the investigator.
* Pregnancy, nursing mother, or unwillingness to use barrier contraception
* Diagnosis of active psychosis, ADHD, ADD
* Current use of medications contraindicated with the use of modafinil-triazolam, Phenobarbital, cyclosporine A, theophylline, carbamazepine, diazepam, phenytoin, mephenytoin, rifampin, ketoconazole, itraconazole,
* Illegal drug or alcohol abuse (defined as two affirmative responses to the CAGE questionnaire)
* Prior use of modafinil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-02; Study Completion 2007-02

PRIMARY OUTCOMES:
Improvement in cognitive efficiency at 6 weeks

SECONDARY OUTCOMES:
Change in performance of cognitive activities at six weeks
Change in fatigue at six weeks
Change in sleep at six weeks
Adverse events, including an increase in SLE activity, at six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J. Harrison, MD, MS, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States